CLINICAL TRIAL: NCT05980598
Title: BelieveIT-201: Phase 2, Randomized Open-labeled Trial of TransCon (TC) TLR7/8 Agonist in Combination With Pembrolizumab or With TC IL-2 β/γ, or Pembrolizumab Alone as Neoadjuvant Therapy for Stage III-IVA Resectable Locoregionally Advanced Head and Neck Squamous Cell Carcinoma
Brief Title: TransCon (TC) TLR7/8 Agonist, TC IL-2 β/γ, Pembrolizumab Prior to Surgery for Advanced Head and Neck Squamous Cell Carcinoma
Acronym: BelieveIT-201
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: The Sponsor made the decision to close enrollment as part of a strategic portfolio review.
Sponsor: Ascendis Pharma A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ASND0038
Record Dates: First submitted 2023-07-20; First posted 2023-08-08 (Actual); Last update posted 2025-08-01 (Actual); Status verified 2025-07

CONDITIONS: Head and Neck Neoplasms
Keywords: HNSCC; Head and Neck Cancer; TransCon TLR7/8 Agonist; TC TLR7/8; TransCon IL-2 β/γ; TC IL-2 β/γ; Neoadjuvant; Neoadjuvant Head and Neck; LA-HNSCC; Locoregionally Advanced HNSCC
MeSH Terms: conditions — Head and Neck Neoplasms; Squamous Cell Carcinoma of Head and Neck | interventions — pembrolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- TransCon TLR7/8 Agonist in combination with pembrolizumab (Experimental): Participants receive 2 cycles, once every 3 weeks of TransCon TLR7/8 Agonist intratumoral (IT) injection in combination with pembrolizumab as a 30-minute intravenous (IV) infusion
  Interventions: Drug: TransCon TLR7/8 Agonist; Drug: Pembrolizumab
- TransCon TLR7/8 Agonist in combination with TransCon IL-2 β/γ (Experimental): Participants receive 2 cycles, once every 3 weeks of TransCon TLR7/8 Agonist (IT injection) in combination with TransCon IL-2 β/γ as a 30-minute IV infusion
  Interventions: Drug: TransCon TLR7/8 Agonist; Drug: TransCon IL-2 β/γ
- Pembrolizumab (Active Comparator): Participants receive 2 cycles, once every 3 weeks of pembrolizumab alone as a 30-minute IV infusion
  Interventions: Drug: Pembrolizumab

INTERVENTIONS:
Drug: TransCon TLR7/8 Agonist — TLR7/8 agonist prodrug
  Arms: TransCon TLR7/8 Agonist in combination with TransCon IL-2 β/γ; TransCon TLR7/8 Agonist in combination with pembrolizumab
Drug: Pembrolizumab — A type of immunotherapy that works by blocking the PD-1 pathway to help prevent cancer cells from hiding
  Other Names: Keytruda™
  Arms: Pembrolizumab; TransCon TLR7/8 Agonist in combination with pembrolizumab
Drug: TransCon IL-2 β/γ — Sustained systemic release of IL-2 β/γ with selective receptor binding that may stimulate the immune system to kill cancer cells
  Arms: TransCon TLR7/8 Agonist in combination with TransCon IL-2 β/γ

SUMMARY:
The purpose of this trial is to evaluate the safety and efficacy of TransCon TLR7/8 Agonist, TransCon IL-2 β/γ, and pembrolizumab given prior to curative intent surgery in treatment of participants with newly diagnosed Stage III/IVA resectable locoregionally advanced head and neck squamous cell carcinoma (LA-HNSCC). After surgery, participants will receive local standard-of-care treatment and will be followed for safety, efficacy, and survival for up to 2 years.

This trial contains a safety run-in to evaluate the safety and tolerability of the two treatment arms: Arm A (TransCon TLR7/8 Agonist plus pembrolizumab) and Arm B (TransCon TLR7/8 Agonist plus TransCon IL-2 β/γ). The safety run-in will be followed by the randomized Phase 2, open-label part of the trial comparing the safety, efficacy and survival of treatment Arm A or Arm B compared to treatment Arm C (pembrolizumab monotherapy).

DETAILED DESCRIPTION:
This is a randomized, Phase 2, open-label, multicenter trial of TransCon TLR7/8 Agonist in combination with pembrolizumab, TransCon TLR7/8 Agonist in combination with TransCon IL-2 β/γ, or pembrolizumab monotherapy as neoadjuvant therapy in participants with Stage III-IVA resectable LA-HNSCC.

This trial starts with a safety run-in of 12 participants, 6 participants each in Arms A (TransCon TLR7/8 Agonist plus pembrolizumab) and B (TransCon TLR7/8 Agonist plus TransCon IL-2 β/γ) randomized 1:1.

After completing the safety run-in, 80 participants will be randomized in a 2:2:1 ratio in 3 treatment Arms A, B or C (pembrolizumab monotherapy).

Once randomized, participants should begin treatment within 5 calendar days. Participants enrolled after the safety run-in, into the 2:2:1 randomization part of the trial, will be stratified as follows: oropharyngeal HPV p16 positive versus oropharyngeal HPV p16 negative or larynx/hypopharyngeal/oral cavity regardless of HPV p16 status. All participants should receive study drug(s) every 21 days (Q21D) for 2 cycles followed by curative-intent surgery. After surgery, participants may receive standard-of-care treatment in the adjuvant setting, as per investigator's decision and local guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Has local histologically confirmed new diagnosis of resectable, non-metastatic, SCC that is either: Stage III tumor HPV-positive oropharyngeal primary that is tumor size (T) 4, lymph node involvement (N) 0-2, no distant metastases (M) 0; Stage III or IVA oropharyngeal tumor HPV-negative; or Stage III or IVA larynx/hypopharynx/oral cavity primaries regardless of HPV status (per American Joint Committee on Cancer [AJCC] Staging, 8th edition).
* Has available archived or fresh core or excisional biopsy of a tumor lesion. Note: Fine needle aspirations may be allowed after discussion with Medical Monitor.
* Is eligible and plans for primary LA-HNSCC surgery based on investigator decision and per local practice.
* Has results from tumor HPV status by p16 immunohistochemistry (IHC) for oropharyngeal tumors. (HPV DNA analysis for HPV tumor status is acceptable if that is the local standard of care analysis.)
* Has adequate organ function at screening.
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1.
* Has at least one lesion that is deemed by the investigator to be easily and safely accessible for IT injection.

Exclusion Criteria:

* Active autoimmune conditions.
* Has significant cardiac disease.
* Has a known bleeding disorder that is deemed to place the participant at unacceptable risk for bleeding complications from IT injections or biopsies.
* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy (in doses exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days prior to randomization.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2023-09-29 (Actual); Primary Completion 2025-03-28 (Actual); Study Completion 2025-03-28 (Actual)

PRIMARY OUTCOMES:
Major Pathological Response | Up to 6 weeks after Cycle 2 (each cycle is 21 days)
  The proportion of participants with a major pathological response (mPR) as assessed by the Central Pathologist at the time of definitive surgery. mPR is defined as ≤10% invasive squamous cell carcinoma within the resected primary tumor specimen and all the sampled regional lymph nodes.

SECONDARY OUTCOMES:
Pathological Complete Response | Up to 6 weeks after Cycle 2 (each cycle is 21 days)
  A central pathology laboratory and local hospital pathologist will evaluate if all the tumor is completely gone from the primary tumor and all the lymph nodes that were removed at surgery.
Event Free Survival | Up to 5 years
  The time from the date of randomization to the date of first record of any of the following events: disease progression; local or distant recurrence determined by radiology scans or tumor biopsy as needed, or death due to any cause.
Overall Survival | Up to 5 years
  The time from randomization to death due to any cause.
Safety and Tolerability | From time of signing of the ICF up to 100 (±7) days following the last dose of study drug
  Incidence and severity of adverse events (AEs) and serious adverse events (SAEs).

CONTACTS AND LOCATIONS:
Overall Officials: Joan Morris, Study Director — Ascendis Pharma Oncology Division A/S
Locations (55):
- United States (16):
  - Ascendis Investigational Site, Los Angeles, California
  - Ascendis Investigational Site, San Francisco, California
  - Ascendis Investigational Site, Chicago, Illinois
  - Ascendis Investigational Site, Springfield, Illinois
  - Ascendis Investigational Site, Iowa City, Iowa
  - Ascendis Investigational Site, Louisville, Kentucky
  - Ascendis Investigational Site, Boston, Massachusetts
  - Ascendis Investigational Site, Detroit, Michigan
  - Ascendis Investigational Site, Rochester, Minnesota
  - Ascendis Investigational Site, New York, New York
  - Ascendis Pharma Investigational Site, Canton, Ohio
  - Ascendis Investigational Site, Cincinnati, Ohio
  - Ascendis Investigational Site, Columbus, Ohio
  - Ascendis Investigational Site, Charleston, South Carolina
  - Ascendis Investigational Site, Knoxville, Tennessee
  - Ascendis Investigational Site, Houston, Texas
- Georgia (3):
  - Ascendis Investigational Site, Kutaisi, Imereti
  - Ascendis Investigational Site, Tbilisi
  - Ascendis Investigational Site II, Tbilisi
- Germany (6):
  - Ascendis Investigational Site, Erlangen, Bavaria
  - Ascendis Investigational Site, Greifswald
  - Ascendis Investigational Site, Jena
  - Ascendis Investigational Site, Leipzig
  - Ascendis Investigational Site, Mannheim
  - Ascendis Investigational Site, Ulm
- Hungary (5):
  - Ascendis Investigational Site, Pécs, Baranya
  - Ascendis Investigational Site, Budapest
  - Ascendis Investigational Site, Debrecen
  - Ascendis Investigational Site, Győr
  - Ascendis Investigational Site, Zalaegerszeg
- Italy (7):
  - Ascendis Investigational Site, Meldola
  - Ascendis Investigational Site, Milan
  - Ascendis Investigational Site, Modena
  - Ascendis Investigational Site, Naples
  - Ascendis Investigational Site, Novara
  - Ascendis Investigational Site, Pavia
  - Ascendis Investigational Site, Rozzano
- Poland (3):
  - Ascendis Investigational Site, Gliwice
  - Ascendis Investigational Site, Siedlce
  - Ascendis Investigational Site, Warsaw
- Spain (11):
  - Ascendis Investigational Site, Barcelona
  - Ascendis Investigational Site, El Palmar
  - Ascendis Investigational Site, L'Hospitalet de Llobregat
  - Ascendis Investigational Site, Lugo
  - Ascendis Investigational Site, Madrid
  - Ascendis Investigational Site II, Madrid
  - Ascendis Investigational Site, Málaga
  - Ascendis Investigational Site, Pamplona
  - Ascendis Investigational Site, Terrassa
  - Ascendis Investigational Site, Valencia
  - Ascendis Investigational Site, Zaragoza
- Taiwan (4):
  - Ascendis Investigational Site, Kaohsiung City
  - Ascendis Investigational Site, Taichung
  - Ascendis Investigational Site, Tainan
  - Ascendis Investigational Site, Taoyuan District

IPD SHARING:
Plan to Share IPD: No